CLINICAL TRIAL: NCT03473132
Title: Assessment of Coagulation Factor Levels in LVAD Patients Following Temporary Warfarin Reversal With 4F-PCC
Brief Title: Assessment of Coagulation Factor Levels in Left Ventricular Device (LVAD )Patients Following Temporary Warfarin Reversal With Four Factor Prothrombin Complex Concentrate (4F-PCC)
Acronym: KVAD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Principal Investigator, Jean M Connors, Director, Hemostatic and Antithrombotic Stewardship Program, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017P001254
Record Dates: First submitted 2018-02-07; First posted 2018-03-22 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Anticoagulation; Anticoagulation Reversal

STUDY DESIGN:
Intervention Model Description: Pilot study of consecutive patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Based on starting international normalized ratio (INR) and target INR, the dose of four factor prothrombin complex concentrate will be calculated and infused. Coagulation factor levels will be assessed over 48-72 hours.
  Interventions: Drug: four factor prothrombin complex concentrate

INTERVENTIONS:
Drug: four factor prothrombin complex concentrate — After treatment with 4F-PCC, coagulation factor levels will be assessed. Time to return to anticoagulation target INR will also be determined.

SUMMARY:
Prospective assessment of vitamin K dependent coagulation factor levels after temporary warfarin reversal in participants with left ventricular assist devices (LAVD).

DETAILED DESCRIPTION:
Prospective evaluation of the levels of the vitamin K dependent coagulation factors 2,7,9,10, and proteins C and S, in patients on warfarin treated with four factor prothrombin complex concentrate (4F-PCC). Participants on vitamin K antagonists (VKA) such as warfarin have suppressed levels that are brought to the normal range with treatment with 4F-PCC to reverse the warfarin effect. The investigators will assess the duration of effect of 4F-PCC on these factor levels in participants with left ventricular assist devices (VAD) requiring temporary reversal of warfarin for invasive procedures that have a risk of bleeding. The investigators will also assess the time to return to therapeutic INR..

ELIGIBILITY:
Inclusion Criteria:

* LVAD on warfarin requiring temporary interruption of anticoagulation for procedures

Exclusion Criteria:

* recent thrombotic event

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-03-15 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
plasma concentration of factors II,VII, IX, X, proteins S and C every 6 hours for 48 hours after treatment with 4F-PCC and correlation with international normalized ratio | through 48 hours
  assessment of change in vitamin K dependent coagulation factor levels after infusion of 4F-PCC

SECONDARY OUTCOMES:
Adverse events | 30 days
  bleeding
adverse events | 30 days
  thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Jean M Connors, MD, Principal Investigator — Brigham and Women';s Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
yes